CLINICAL TRIAL: NCT07153913
Title: Comprehensive Nutritional Support for Children in Zambia (ZamCNC) - A Pilot Investigation
Acronym: ZamCnC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Günther Fink (Other)
Responsible Party: Sponsor-Investigator, Günther Fink, Unit Head and Professor, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZamCnC
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Malnourished Children; Stunting of Growth
Keywords: stunting; food supplementation; counseling; cash tranfers
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Families in control group will not receive any support through the study
- Food provision and nutritional counseling (Experimental): Families will receive intensive support including bi-weekly nutritional counseling and weekly dropoffs of locally acquired food.
  Interventions: Other: Intensive growth support

INTERVENTIONS:
Other: Intensive growth support — For women in the intervention group, we will develop a nutritional plan for the child in collaboration with the mother. Mothers will then receive a visit every other week - during this visit, children's health and nutrition will be discussed, and height and weight will be measured by field officers. Detailed food recommendations will be made based on national and international infant and young child feeding guidelines. To ensure appropriate foods are available, field workers will drop off local foods on a weekly basis.
  Arms: Food provision and nutritional counseling

SUMMARY:
In a recently completed intervention study, more than 50% of children in Lusaka were found to be stunted by age two, even when nutritional supplements were provided. It seems likely that these high rates of stunting are primarily due to inadequate basic nutritional intake. The main goal of this project is investigate this conjecture through a small pilot study that will be conducted in the urban area of Lusaka.

DETAILED DESCRIPTION:
This is very small cluster-randomized trial, with 64 families recruited from 4 selected neighbourhoods. 2 of these neighbourhoods will be selected for nutritional counselling and food support.

Children ages 6-12 months old and their caregivers will be included. Exclusion criteria: low birth weight; planning to move; twins.

All families will complete a baseline and endline assessment - each lasting approximately 30-45 minutes.

Children in the two intervention clusters will receive a visit every two weeks to discuss child nutrition, and to monitor height and weight gains. We will also provide additional food/groceries to mothers in the treatment group, i.e. to the 32 families in the two neighborhoods selected for treatment.

ELIGIBILITY:
Inclusion Criteria:Only children who are 6-12 months old at the time of recruitment and their caregivers in selected areas will be eligible for the study.

Exclusion Criteria:

* expected to move
* no child health card
* participating in cash transfer programs

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Height-for-age z-score | measured approximately 6 months after initiation of intervention
  Children's height for age z-score after six months of interventions

CONTACTS AND LOCATIONS:
Overall Officials: Günther Fink, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Innovations for Poverty Action Zambia, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: No